CLINICAL TRIAL: NCT02406768
Title: The Neurodevelopment in Normal Children in Cambodia and Thailand
Brief Title: A Sub-study of PREDICT Neurodevelopment Protocol
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 035.4
Record Dates: First submitted 2014-03-31; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Neurocognitive Development
Keywords: normal controls

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV negative unexposed: HIV negative controls
- HIV negative exposed: HIV-negative children born to HIV-infected mothers

SUMMARY:
To determine the neurodevelopment (ND) in normal children in Thailand and Cambodia and to use this group to compare the neurodevelopmental changes over time to the HIV-infected children with and without HAART (main study).

DETAILED DESCRIPTION:
Normative data are mostly, if not exclusively, obtained from children in the Western world. Comparing data from Asian children to these norms may lead to the wrong interpretation of the results, as it does not account for cultural differences, translation issues and a possibly different education system. Therefore it is essential to include a matched control group to evaluate the participants of the study to the fullest extent in terms of cognition, memory, behavior and fine motor skills, in all age groups over the full course of the study.

ELIGIBILITY:
Inclusion Criteria: for HIV negative exposed children

* Child from a HIV-positive mother
* Documented negative test for HIV-1 infection
* Between the age from 1-15 years
* Caregiver of the subject is willing and able to sign informed consent, prior to the study
* Thai or Cambodian origin

HIV negative and not HIV exposed:

Inclusion

* Child from a HIV-negative mother (by history)
* Documented negative test for HIV-1 infection
* Between the age from 1-15 years
* Caregiver of the subject is willing and able to sign informed consent, prior to the study
* Thai or Cambodian origin

Exclusion Criteria: for HIV negative exposed children

* The inability of the caregivers to understand the nature and extend of the trial and the procedure required
* Patients with psychiatric disorder
* Patients with a syndrome that affects cognitive performance

for HIV negative and not HIV exposed

* The inability of the caregivers to understand the nature and extent of the trial and the procedure required
* Patients with psychiatric disorder
* Patients with a syndrome that affects cognitive performance

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: HIV negative unexposed and HIV-negative children born to HIV-infected mothers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
neurodevelopment changes (composite of cognitive, fine motor and behavioral) | up to 96 weeks
  measured by cognitive test, fine motor test and behavioral assessment test

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (10):
- Cambodia (2):
  - National Center for HIV/AIDS, Dermatology and STDs (NCHADS), Phnom Penh
  - National Pediatric Hospital, Phnom Penh
- Thailand (8):
  - Pediatric Infectious Diseases Unit Department of Pediatrics Faculty of Medicine Chulalongkorn University, Bangkok, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), The Thai Red Cross AIDS Research Center, Bangkok, Bangkok
  - Prapokklao Hospital, Chanthaburi, Changwat Chanthaburi
  - Chiangrai Regional Hospital, Chiang Rai, Changwat Chiang Rai
  - Queen Savang Vadhana Memorial Hospital, Pediatric Department,, Chon Buri, Changwat Chon Buri
  - Department of Pediatrics Faculty of Medicine Khon Kaen University, Khon Kaen, Changwat Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi, Changwat Nonthaburi
  - Nakornping Hospital, Chiang Mai, Chiang Mai

REFERENCES:
- [Result] Puthanakit T, Ananworanich J, Vonthanak S, Kosalaraksa P, Hansudewechakul R, van der Lugt J, Kerr SJ, Kanjanavanit S, Ngampiyaskul C, Wongsawat J, Luesomboon W, Vibol U, Pruksakaew K, Suwarnlerk T, Apornpong T, Ratanadilok K, Paul R, Mofenson LM, Fox L, Valcour V, Brouwers P, Ruxrungtham K; PREDICT Study Group. Cognitive function and neurodevelopmental outcomes in HIV-infected Children older than 1 year of age randomized to early versus deferred antiretroviral therapy: the PREDICT neurodevelopmental study. Pediatr Infect Dis J. 2013 May;32(5):501-8. doi: 10.1097/INF.0b013e31827fb19d. PMID 23263176
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org